CLINICAL TRIAL: NCT02810548
Title: Clinical and Biochemical Evaluation of Platelets Rich Fibrin (PRF) and Nanohydroxyapatite in the Treatment of Intrabony Defects
Brief Title: Evaluation of Platelets Rich Fibrin and Nanohydroxyapatite in the Treatment of Intrabony Defects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maha A. Bahammam, Associate Professor and Consultant of Periodontology, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 032-16
Record Dates: First submitted 2016-06-08; First posted 2016-06-23 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Bony Defects
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- OFD alone (Placebo Comparator): Control group: including 15 defects that will receive open flap debridement (OFD).
  Interventions: Procedure: OFD alone
- PRF + OFD (Active Comparator): Test group (1): including 15 defects that will receive platelet rich fibrin (PRF) with open flap debridement (OFD).
  Interventions: Procedure: OFD alone; Drug: Platelet rich Fibrin
- Bone + OFD (Active Comparator): Test group (2): including 15 defects that will receive nanohydroxyapatite bone graft with open flap debridement OFD).
  Interventions: Procedure: OFD alone; Drug: Nanohydroxyapatite
- PRF + Bone + OFD (Active Comparator): Test group (3): including 15 defects that will receive nanohydroxyapatite bone graft with platelet rich fibrin (PRF) after open flap debridement (OFD).
  Interventions: Procedure: OFD alone; Drug: Platelet rich Fibrin; Drug: Nanohydroxyapatite

INTERVENTIONS:
Procedure: OFD alone — Periodontal surgical cleaning procedure
  Other Names: Periodontal Surgery
Drug: Platelet rich Fibrin — Natural platelet concentrate rich in growth factors
  Other Names: Natural growth factor
  Arms: PRF + Bone + OFD; PRF + OFD
Drug: Nanohydroxyapatite — Synthetic bone graft
  Other Names: Bone graft
  Arms: Bone + OFD; PRF + Bone + OFD

SUMMARY:
Background: the ultimate goal of periodontal therapy is the regeneration of periodontal tissues. Researches had demonstrated the benefits of platelet concentrates bine grafts in osseous regeneration in the areas of periodontal surgery.

Aim of the study: to evaluate the effect of PRF with/without nanohydroxyapatite in periodontal intrabony defects.

DETAILED DESCRIPTION:
Background: the ultimate goal of periodontal therapy is the regeneration of periodontal tissues. The regenerative and wound healing potential of platelets has attracted much attention over the last few years. Researches had demonstrated the benefits of platelet concentrates in osseous regeneration in the areas of periodontal surgery and implantology. In addition, nanohydroxyapatite was shown to be unsheathed by newly formed bone and partly replaced by it, but resorbed very slowly, as shown in animal experiments after 9 months or in clinical studies after a 6-month observation period. The clinical and biochemical studies evaluating the regenerative effect of PRF alone or in combination with nanohydroxyapatite in periodontal intrabony defects are still deficient.

Aim of the study: to evaluate clinical and biochemical effect of PRF with/without nanohydroxyapatite in treatment of human intrabony defects.

ELIGIBILITY:
Inclusion Criteria:

* All patients are free from systemic illness.
* All patients should be diagnosed as having chronic periodontitis.
* Patients should be cooperative, motivated and willing to follow our treatment protocol and follow up visits.
* Patients selected had not received antibiotics or anti-inflammatory therapy in the 6 months prior to examination.

Exclusion Criteria:

* Presence of areas of periodontal pocket of (probing depth ≥5 and clinical attachment level (CAL) ≥ 3).
* Patients who have received any type of periodontal treatment in the past 6 months prior to examination.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in Gingival crevicular fluid (GCF) | up to 3 weeks.
  GCF will be collected after removing saliva and supra-gingival plaque using methylcellulose filter paper strip that will be inserted in the periodontal pocket and will be let in for 30 seconds.

SECONDARY OUTCOMES:
Changes in Gingival index | up to 3 months
  Gingival index (GI) developed on 1963.
Changes in level of attachment loss | up to 3 months
  Attachment loss: will be measured from the cemento-enamel junction (CEJ) to the apical part of the sulcus.
Changes in probing pocket depth | up to 3 months
  Probing pocket depth (PD): six measurements per tooth will be recorded by using the University of Michigan O periodontal probe with Williams markings.

CONTACTS AND LOCATIONS:
Overall Officials: Maha A Bahammam, DSc, Principal Investigator — King Abdelaziz University
Locations (1):
- King Abdelaziz University. Faculty of dentistry, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No